CLINICAL TRIAL: NCT01726504
Title: The Efficacy and Safety Study of Electro-acupuncture for Severe Chronic Functional Constipation - a Multi-center, Randomized Controlled Trial
Brief Title: The Efficacy and Safety Study of Electro-acupuncture for Severe Chronic Functional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Liu Baoyan, Vice President of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012BAI24B01
Record Dates: First submitted 2012-10-30; First posted 2012-11-15 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Constipation
Keywords: chronic functional constipation; electro-acupuncture; multi-center randomized controlled trial; efficacy; safety
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- electro-acupuncture (Experimental): 1. The electric stimulator is applied to bilateral ST25andSP14 with dilatational wave10/50 Hz and electric current0.1-1.0mA.They are given acupuncture with 0.3×50mm or 0.35×75mm needles by inserting30-70mm and twirling lifting andthrusting 3 times.Dosage:The needle arrives the abdominal muscle layer(patients feel painful and acupuncturists feel touching hard).
  2. Bilateral ST37 are given conventional acupuncture with 0.30mm×40mm needles by inserting 25-30mm and twirling lifting and thrusting for 3.Dosage:Local sour and heavy feeling is the appropriate dose.
  Every session lasts for 30min/day.The participants are treated continuously for 8 weeks.During 8-week treatment the first 2 weeks,5 sessions per week,and 3 sessions per week in the rest 6 weeks,28 sessions for each patients in total.
  Interventions: Device: electro-acupuncture
- sham electro-acupuncture (Sham Comparator): 1. The electric stimulator is applied to bilateral sham ST25 and sham SP14 with dilatational wave, 10/50 Hz and electric current 0.5mA. The mental wire has been cut off with a same outlook as the treatment group. The electric stimulator is looked normal but with no current output. The needle is inserted by 3mm-5mm (the needle can be vertically fixed on the skin).
  2. Bilateral ST37 are given acupuncture with 3mm-5mm (the needle can be vertically fixed on the skin).
  Length of Treatment and the treatment sessions are the same as treatment group.
  Interventions: Device: sham electro-acupuncture

INTERVENTIONS:
Device: electro-acupuncture — Procedure: electro-acupuncture; Points:Tianshu (ST25) Fujie(SP14), Shangjuxu (ST37).Pierced the skin, needles are inserted 30to70mm into bilateral ST25 and SP14 vertically until piercing the abdominal muscle layer.Electric stimulator is applied to bilateral ST25 and SP14 with dilatational wave, 10/50 Hz and electric current 0.1-1.0mA. The participant's abdominal muscle twitching mildly is the appropriate dose. Bilateral ST37 are inserted 25-30mm and then twirling lifting and thrusting for 3 times.Local sour and heavy feeling is appropriate dose. Steady small twirling lifting and thrusting 3 times in all. 30 min/per day/per session.During the 8 weeks treatment, the first 2 weeks,5 sessions per week, and 3 sessions per week in the rest 6 weeks,28 sessions for each patients in total.
  Other Names: SDZ-V electro-acupuncture apparatus (Huatuo, made in China)
  Arms: electro-acupuncture
Device: sham electro-acupuncture — Procedure:sham electro-acupuncture;Points:Sham Tianshu(ST25),sham Fujie(SP14),sham Shangjuxu (ST37).Sham points location:20mm away from ST25,middle of Spleen and Stomach Channel;30mm from SP14,middle of Spleen and Stomach Channel; one point beside ST37,middle of Stomach and Gallbladder Channel; Performance:The needle is inserted with needle of 0.30×25mm by 3-5mm. No twirling lifting and thrusting. The electric stimulator is applied to bilateral sham ST25 and sham SP14 with dilatational wave,10/50 Hz and electric current 0.5mA.The mental wire has been cut off with a same outlook as the treatment group.The electric stimulator is looked normal but with no current output. Length of Treatment and the treatment sessions are the same as treatment group.
  Other Names: Sham SDZ-V electro-acupuncture apparatus (Huatuo, China)
  Arms: sham electro-acupuncture

SUMMARY:
The main purpose of this study is to evaluate efficacy of electro-acupuncture for severe functional constipation compared with sham acupuncture, used as placebo; the secondary purpose is to evaluate the safety and post-treatment effect of electro-acupuncture.

DETAILED DESCRIPTION:
Chronic functional constipation is a common disease. To date there has not specific therapy on chronic functional constipation. Systematic reviews indicate that acupuncture is probably effective for the disease, but the evidence is limited. Recently, we have finished a multi-center clinical trial of individualized deep electro-acupuncture (EA) for chronic functional constipation (n=460, Registration ID: NCT00508482) which preliminarily showed EA was effective.

This multi-center large-sample randomized controlled clinical trial of acupuncture for severe functional constipation is designed to confirm the efficacy and safety of EA.

This project is conducted by Chinese experts, supported by the Chinese Government. The research result is expected to provide high quality evidence of EA for chronic functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* meeting the diagnosis of Rome III criteria for chronic functional constipation;
* severe chronic constipation: two or fewer spontaneous complete bowel movements per week for more than 3 months;
* 18-75 years old;
* no use of medicine for constipation during the two weeks before enrollment (except rescue medication);
* no acupuncture treatment for constipation in recent 3 months;
* never joined any other trial in process in 3 months;
* volunteered to join this research and signed the informed consent.

Exclusion Criteria:

* Irritable bowel syndrome (IBS) and constipation caused by endocrine, metabolic, nervous or postoperative diseases or drugs;
* constipation accompanied by serious cardiovascular, hepatic, renal, or psychiatric disease, cognitive dysfunction or aphasia, or severe dystrophy affecting the cooperation for examination or treatment;
* pregnant women or women in lactation period
* constipation accompanied by abdominal aneurysm, hepatosplenomegaly, etcetera;
* bleeding disorders, or regular anticoagulant drug users, such as warfarin and heparin, etcetera;
* cardiac pacemaker carrier.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1075 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baoyan Liu, Master, Principal Investigator — Vice President of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang Y, Liu Y, Zhou K, Bauer BA, Liu B, Su T, Mo Q, Liu Z. The duration of acupuncture effects and its associated factors in chronic severe functional constipation: secondary analysis of a randomized controlled trial. Therap Adv Gastroenterol. 2019 Oct 9;12:1756284819881859. doi: 10.1177/1756284819881859. eCollection 2019. PMID 31636713
- [Derived] Liu Z, Yan S, Wu J, He L, Li N, Dong G, Fang J, Fu W, Fu L, Sun J, Wang L, Wang S, Yang J, Zhang H, Zhang J, Zhao J, Zhou W, Zhou Z, Ai Y, Zhou K, Liu J, Xu H, Cai Y, Liu B. Acupuncture for Chronic Severe Functional Constipation: A Randomized Trial. Ann Intern Med. 2016 Dec 6;165(11):761-769. doi: 10.7326/M15-3118. Epub 2016 Sep 13. PMID 27618593
- [Derived] Liu Z, Liu J, Zhao Y, Cai Y, He L, Xu H, Zhou X, Yan S, Lao L, Liu B. The efficacy and safety study of electro-acupuncture for severe chronic functional constipation: study protocol for a multicenter, randomized, controlled trial. Trials. 2013 Jun 15;14:176. doi: 10.1186/1745-6215-14-176. PMID 23768191

RESULTS

PARTICIPANT FLOW:
Groups:
- Electro-acupuncture: The acupuncture points are ST25, SP14,ST37. After sterilizing the skin, filiform needles are inserted 3 to 8 cm into bilateral ST25 and SP14 vertically and slowly without any manipulation until arrive the abdominal muscle layer(patients feel painful and acupuncturists feel touching hard). An electric stimulator (SDZ-V EA apparatus; Huatuo, China) is applied to bilateral ST25 and SP14 with a dilatational wave of 10/50 Hz and electric current between 0.1 and 1.0 mA with abdominal muscle twitching mildly indicating the appropriate dose.
  The bilateral ST37 is inserted 3cm - twirling, lifting and thrusting three times. A local sour and heavy feeling indicates the appropriate dose.
  Every session lasts for 30min/day. The participants are treated continuously for 8 weeks. During 8-week treatment the first 2 weeks,5 sessions per week, and 3 sessions per week in the rest 6 weeks,28 sessions for each patients in total.
- Sham Electro-acupuncture: The acupuncture points are sham ST25, SP14, ST37. Sham location points are: about 2cm away from ST25,in the middle of the spleen and stomach channel; about 3 cm from SP14, in the middle of the spleen and stomach channel; one point beside ST37, in the middle of the stomach and gallbladder channel. The needle is inserted after sterilizing the skin by 1 to 1.5 cm, until the needle can be vertically fixed on the skin. No twirling lifting and thrusting manipulation is used. The sham electric stimulator (sham SDZ-V EA apparatus; Huatuo) is applied to the bilateral sham ST25 and sham SP14 with a dilatational wave of 10/50 Hz and electric current of 0.5 mA. The metal wire has been cut off inside to give the appearance of the real electric stimulator, with no current output. Length of treatment and the treatment sessions are the same as the treatment group sessions are the same as the treatment group.
Period: Overall Study
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Started | 536 | 539
Completed | 524 | 511
Not Completed | 12 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture | Total
Number analyzed (Participants) | 536 | 539 | 1075
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 447 | 457 | 904
  >=65 years | 89 | 82 | 171
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 415 | 407 | 822
  Male | 121 | 132 | 253
Race/Ethnicity, Customized [Number; unit: participants]
  Han | 519 | 526 | 1045
  Man | 5 | 2 | 7
  Hui | 8 | 9 | 17
  Zhuang | 1 | 2 | 3
  Miao | 0 | 0 | 0
  Wei | 0 | 0 | 0
  other | 3 | 0 | 3
Body-mass index [Mean (Standard Deviation); unit: kg/m^2] — Body-mass index was measured by research assistants.Data were tested using Student's t test.
  kg/m^2 | 22.32 (3.04) | 22.75 (3.00) | 22.54 (3.03)
Constipation duration (mon) [Mean (Standard Deviation); unit: month] — Constipation duration was self-reported by participants.Data were tested using Student's t test.
  month | 130.81 (122.61) | 132.71 (127.00) | 131.76 (124.78)
Coexisting illness [Number; unit: participants] — Coexisting illnesses was self-reported by participants.Data were tested using chi-square test.
  participants
    Diabetes | 11 | 10 | 21
    Hypertension | 41 | 39 | 80
    Digestive system disease | 11 | 16 | 27
    Others | 78 | 71 | 149
    None | 395 | 403 | 798
Use of Other Measures by Participants [Number; unit: participants] — Use of Other Measures by Participants:Data were tested using chi-square test.
  participants
    Rescue medicine | 170 | 147 | 317
    Others | 17 | 19 | 36
    None | 349 | 373 | 722
average number of times other measures were used [Mean (Standard Deviation); unit: number of times per week] — Average number of times other measures were used self-reported by participants.Data were tested using Student's t test.
  number of times per week
    Rescue medicine | 0.66 (1.47) | 0.62 (1.91) | 0.64 (1.71)
    Others | 0.08 (0.58) | 0.06 (0.43) | 0.07 (0.51)
Complete Spontaneous Bowel Movements (CSBMs) Per Week [Mean (Standard Deviation); unit: number of times] — Number of CSBMs/week during the 2-week screening period was calculated from participants' diaries by summing weekly CSBMs or SBMs then dividing by two.Data were tested using Student's t test.
  number of times | 0.39 (0.62) | 0.42 (0.62) | 0.41 (0.62)
Spontaneous Bowel Movements (CSBMs) Per Week [Mean (Standard Deviation); unit: number of times] — SBMs/week during the 2-week screening period was calculated from participants' diaries by summing weekly CSBMs or SBMs then dividing by two.
  number of times | 1.90 (1.34) | 2.02 (1.45) | 1.96 (1.40)
Score of Patient Assessment of Constipation Quality of Life(PAC-QOL) [Mean (Standard Deviation); unit: scores on a scale] — The PAC-QOL was administered by research assistants at the baseline visit and was reported by participants.Data were tested using Student's t test.PAC-QOL scale ranges are 28-140,and higher values represent a worse outcome.Subscales are summed to compute the total score.
  scores on a scale | 77.06 (19.27) | 75.06 (19.26) | 76.06 (19.28)

OUTCOME MEASURES:

1. Primary Outcome: the Change in Mean Weekly CSBMs During Weeks 1-8 Since Treatment
Description: the change number in mean weekly CSBMs during weeks 1-8 since treatment compared with baseline.
Time Frame: Baseline and weeks 1-8
Measure: Mean (Standard Error); unit: number of times
Groups:
- Electro-acupuncture: Electroacupuncture (EA) group consisted of 28 sessions of 30 minutes' duration, each administered over a period of 8 weeks. Huatuo disposable needles and EA apparatus, type SDZ-V(Suzhou Medical Appliance, China) were used. Participants in the EA group received EA at bilateral acupoints of ST25, SP14,ST37. With participant supine, 0.30 mm×50 mm or 0.35mm×75mm needles were inserted into ST25 and SP14 slowly and vertically, without manipulation, for approximately 30 to 70mm until they pierced the muscle layer of the abdominal wall. EA apparatus were attached transversely to bilateral ST25 and SP14, lasted for 30 minutes with a dilatational wave of 10/50Hz and current intensity of 0.1 to 1 mA depending on participant's comfort level. 0.30mm × 40mm needles were inserted into ST37 vertically for about 30mm and three small, equal manipulations of twirling, lifting, and thrusting were performed to reach acupuncture de qi.
- Sham Electro-acupuncture: Sham Electroacupuncture (SA) group consisted of 28 sessions of 30 minutes' duration, each administered over a period of 8 weeks (five sessions in each of the first 2 weeks, followed by 3 sessions per week in the remaining 6 weeks). Huatuo disposable needles and EA apparatus, type SDZ-V (Suzhou Medical Appliance, China) were used. Participants in SA group received needling at bilateral non-acupoints of sham ST25, sham SP14, sham ST37. Specifically, 0.30 mm × 25 mm needles were used to penetrate the skin vertically at approximately 3 to 5 mm without any manipulation. Similar to EA group, paired alligator clips from the specially constructed EA apparatus were attached to the needle holders. When switched on, the EA apparatus in the SA group had the same working power indicator and sound but no actual current output. Additionally, 0.30 mm × 25 mm needles were inserted into sham ST37 vertically at about 3 - 5 mm without manipulation.
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Number analyzed (Participants) | 536 | 539
number of times | 1.72 (0.12) | 0.82 (0.13)
Statistical Analysis 1: Comparison: Electro-acupuncture vs Sham Electro-acupuncture; During the 8-week treatment period, the adjusted change from baseline in mean weekly CSBMs was 1.72 ± 0.12 (95% CI, 1.48 to 1.96) in the EA group and 0.82 ± 0.13 (95% CI, 0.58 to 1.07, P<0.001) times more than that in the SA group; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

2. Secondary Outcome: the Percentage of Participants With Three or More Weekly CSBMs
Description: the percentage of participants with three or more weekly CSBMs during weeks 1-8 and weeks 9-20
Time Frame: 1-20 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Number analyzed (Participants) | 536 | 539
percentage of participants
  Week 1-8 | 31.34 | 12.06
  Week 9-20 | 37.69 | 14.10

3. Secondary Outcome: Changes in Mean Weekly CSBMs During Weeks 9-20
Description: The changed number in mean weekly average CSBMs during 9-20th weeks, compared with baseline.
Time Frame: Baseline and weeks 9-20
Measure: Mean (Standard Error); unit: number of times
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Number analyzed (Participants) | 536 | 539
number of times | 1.93 (0.14) | 0.82 (0.14)

4. Secondary Outcome: Mean Weekly SBMs During Weeks 1-8
Description: The changed number in mean of weekly average SBMs (spontaneous bowel movement) during 8-week treatment, compared with baseline.
Time Frame: Baseline and weeks 1-8
Measure: Mean (Standard Error); unit: number of times
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Number analyzed (Participants) | 536 | 539
number of times | 2.30 (0.10) | 1.28 (0.10)

5. Secondary Outcome: Mean Scores for Stool Consistency and Straining During Weeks 1-8
Description: average weekly stool consistency (Bristol Stool Scale) assessment of self-defecation during the 1-8weeks of treatment,compared with baseline. Bristol Stool Scale including 7-type, scored by 1 to 7 respectively.Type 1: Separate hard lumps, like nuts (hard to pass); Type 2: Sausage-shaped, but lumpy; Type 3: Like a sausage but with cracks on its surface; Type 4: Like a sausage or snake, smooth and soft; Type 5: Soft blobs with clear cut edges (passed easily); Type 6: Fluffy pieces with ragged edges, a mushy stool; Type 7: Watery, no solid pieces. Entirely liquid. Type 3, 4 are normal.
Time Frame: Baseline and weeks 1-8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Number analyzed (Participants) | 536 | 539
score on a scale | 0.87 (0.05) | 0.62 (0.04)

6. Secondary Outcome: Change of Average Weekly Degree of Difficulty in Defecation From Baseline
Description: The degree of straining during self-defecation: The severity of straining is graded using a 4-point ordinal scale.
  0 = not at all
  1. = more straining than not
  2. = a great deal
  3. = an extreme amount, need finger manipulation to defecate average weekly degree of difficulty in self-defecation during 1-8weeks,compared with baseline
Time Frame: Baseline and weeks 1-8
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Number analyzed (Participants) | 536 | 539
scores on a scale | -0.74 (0.03) | -0.52 (0.03)

7. Secondary Outcome: Then Change Score of Health-related Quality of Life Via Patient-Assessment of Constipation Quality Of Life (PAC-QOL)
Description: Patient-Assessment of Constipation Quality Of Life(PAC-QOL) ranges are 28-140,and higher values represent a worse outcome.Subscales are summed to compute the total score. The changed score of PAC-QOL at week 8, compared with baseline.
Time Frame: baseline and the end of 8th week
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Number analyzed (Participants) | 536 | 539
score on a scale | -25.65 (2.39) | -18.21 (2.39)

8. Secondary Outcome: Number of Participants With Adverse Events Related to Acupuncture
Time Frame: 1-8 weeks
Measure: Number; unit: participants
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Number analyzed (Participants) | 536 | 539
participants | 31 | 24

9. Secondary Outcome: Mean of Weekly Frequency of Rescue Medicine and Other Defecation Assistances Used
Description: Rescue medicine for constipation during the trial will be recorded. For rescue medicine, any participants experiencing no bowel movements for 3 or more consecutive days during the whole trial period were allowed to use a 110 ml glycerol anal enema or 40-60 ml sorbitol anal enema as a rescue medicine with documentation in the stool diary.Other If a patient used other medicine, it should be also recorded in the diary.Only the frequences of rescue medicine and other medicine for constipation will be recorded in diary by patient. Weekly frequencies were combined across Weeks 1-8 and 9-20 per participant by averaged across all measurements.
Time Frame: 1-20 weeks
Measure: Mean (Standard Error); unit: number of times per week
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Number analyzed (Participants) | 536 | 539
number of times per week
  Week 1-8：Rescue medicine | 0.34 (0.04) | 0.52 (0.06)
  Week 1-8：others | 0.02 (0.01) | 0.02 (0.01)
  Week9-20：Rescue medicine | 0.25 (0.04) | 0.37 (0.05)
  Week 9-20：others | 0.02 (0.01) | 0.06 (0.02)

10. Secondary Outcome: The Number of Participants Using Rescue Medicine for Constipation
Time Frame: 1-20 weeks
Measure: Number; unit: participants
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Number analyzed (Participants) | 536 | 539
participants
  Week 1-8：Rescue medicine | 155 | 183
  Week 1-8：others | 15 | 17
  Week9-20：Rescue medicine | 104 | 124
  Week 9-20：others | 12 | 17

11. Secondary Outcome: Percentage of Weekly Frequency of Rescue Medicine and Other Defecation Assistances Used
Description: as for outcome 9
Time Frame: 1-20 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Number analyzed (Participants) | 536 | 539
percentage of participants
  Week 1-8：Rescue medicine | 28.92 | 33.95
  Week 1-8：others | 2.8 | 3.15
  Week9-20：Rescue medicine | 19.40 | 23.01
  Week 9-20：others | 2.24 | 3.15

ADVERSE EVENTS:
Time Frame: All through the study
Description: All Adverse events（AE）were recorded and measured by both participants themselves and acupuncturists.3 cases(2 in electro-acupuncture(EA)group and 1 in sham EA group)dropped out of this research before getting any intervention for effect,only having baseline data.Multipl imputation was adopted for these 3 in outcome measure part,but not for AE part.
Arm/Group | Electro-acupuncture | Sham Electro-acupuncture
Serious Adverse Events (participants affected / at risk) | 0/534 | 0/538
Other Adverse Events (participants affected / at risk) | 31/534 | 24/538
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electro-acupuncture (N=534) | Sham Electro-acupuncture (N=538)
Left needle (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nausea during acupuncture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Faint during acupuncture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Unbearable pricking (VAS≥8) (Injury, poisoning and procedural complications) | 3 (5) | 5 (6)
Pricking lasted more than 0.5 hour (Injury, poisoning and procedural complications) | 2 (5) | 1 (3)
Hematoma around the site of needling (Injury, poisoning and procedural complications) | 19 (40) | 17 (31)
Bleeding/numbness/infection around the site of needling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Sleeplessness after acupuncture (Injury, poisoning and procedural complications) | 1 (27) | 0 (0)
Dizziness after acupuncture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Other discomforts after acupuncture (Injury, poisoning and procedural complications) | 7 (9) | 1 (2)

LIMITATIONS AND CAVEATS:
The 8-week treatment and 12-week follow-up may not be long enough for EA to show its specific therapeutic effect. Efficacy of electro-acupuncture in relieving severe constipation was evaluated without classifying the types of constipation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes